CLINICAL TRIAL: NCT06803277
Title: Evaluation of Post Operative Pain After a Single Session of Endodontic Retreatment Using Different Root Canal Sealers
Brief Title: Post Operative Pain After Endodontic Retreatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Salih DÜZGÜN, Associate Professor, TC Erciyes University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021/306
Record Dates: First submitted 2025-01-17; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Retreatment
Keywords: endodontic retreatment; root canal sealer; post operative pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: a randomized clinical trial
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Epoxy resin based sealer (Other): AH plus
  Interventions: Procedure: endodontic retreatment
- Calcium silicate based sealer (Other): Sureseal
  Interventions: Procedure: endodontic retreatment
- Calcium hydroxide based sealer (Other): Sealapex
  Interventions: Procedure: endodontic retreatment

INTERVENTIONS:
Procedure: endodontic retreatment — Root canal retreatment is recommended when endodontic disease persists or develops after root canal treatment. Root canal retreatment is believed to be the elimination of the main causes of treatment failure.

SUMMARY:
Clinical Trial The aim of this clinical study was to evaluate the effect of different root canal sealers on post operative pain after a single session endodontic retreatment of the teeth have single root and canal with chronic apical periodontitis.

The main questions aimed to be answered are:

Which of the patients treated with AHplus, Sureseal and Sealapex root canal sealers had more postoperative pain after endodontic retreatment?

Which of the patients that treated with AHplus, Sureseal and Sealapex root canal sealers required more analgesic intake after endodontic retreatment?

Participants:

Undergo a single session of endodontic retreatment using one of AH plus, Sureseal or Sealapex root canal sealers.

Visit the clinic one week later after endodontic retreatment Write the condition of analgesic intake and pain score at 6, 12, 24 hours and 2, 3, 4, 5, 6 and 7 days after treatment using a visual analog scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients who did not have any systemic disease, pregnancy or breastfeeding,
* Patients who were older than 18 years,
* Patients who had not used analgesics, anti-inflammatory or antibiotics in the last 7 days and cortisone in the last 6 months,
* Patients who had improved communication skills and were at a mental level to express pain scoring clearly,
* Patients who did not have bruxism problem or primary contact were included in the study.
* Teeth with more than 60% of the root canal filled have preoperatively asymptomatic single root and single canal with previous root canal treatment and chronic apical periodontitis and periapical index (PAI) scores 2-4

Exclusion Criteria:

* Teeth had root resorption,
* Teeth had crown damage
* Teeth had severe malocclusion,
* Teeth had PAI scores 1 and 5
* Immature teeth

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2021-05-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-01-07 (Actual)

PRIMARY OUTCOMES:
the evaluation of post operative pain levels of the participants after used the different root canal sealers during endodontic retreatment endodontic retreatment | Postoperative pain was assessed using a visual analog scale (VAS) at 6 hours,12 hours, 24 hours, 48 hours, 72 hours, 4,5,6 and 7 days after the end of the retreatment.The VAS was a 100 mm horizontal scale with marks every 10 mm
  The time when the retreatment is completed is considered the start time ( 0 h).Postoperative pain was assessed using a VAS at 6 hours,12 hours, 24 hours, 48 hours, 72 hours, 4,5,6 and 7 days after the end of the retreatment.The VAS was a 100 mm horizontal scale with marks every 10 mm and no numbers except a 0 at the beginning of the scale and a 10 at the end.An investigator blinded to the study groups trained all participants to use the scale.The pain levels were classified as no pain (0-4 mm), mild pain (5-44 mm), moderate pain (45-74 mm), or severe pain (75- 100 mm).
the evaluation of analgesic intake of the participants after used the different root canal sealers during endodontic retreatment | Participants were asked to note whether they took 400 mgr ibuprofen at 6 hours,12 hours, 24 hours, 48 hours, 72 hours, 4,5,6 and 7 days after the end of the retreatment as score 1 or score 2
  The time when the retreatment is completed is considered the start time ( 0 h). Score 1: If the participant did not need analgesic a medicine(400 mgr ibuprofen ) after the retreatment, the participant was told to mark a score of 1.
  Score 2: If the participant needed analgesic a medicine (400 mgr ibuprofen ) after the retreatment, the participant was told to mark a score of 2.

CONTACTS AND LOCATIONS:
Overall Officials: Salih DÜZGÜN, Associate Professor, Study Director — TC Erciyes University
Locations (2):
- Turkey (Türkiye) (2):
  - Erciyes University, Melikgazi, Kayseri
  - Erciyes University, Kayseri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gomes-Filho JE, Watanabe S, Cintra LT, Nery MJ, Dezan-Junior E, Queiroz IO, Lodi CS, Basso MD. Effect of MTA-based sealer on the healing of periapical lesions. J Appl Oral Sci. 2013;21(3):235-42. doi: 10.1590/1679-775720130089. PMID 23857649
- [Result] Nosrat A, Dianat O, Verma P, Nixdorf DR, Law AS. Postoperative Pain: An Analysis on Evolution of Research in Half-Century. J Endod. 2021 Mar;47(3):358-365. doi: 10.1016/j.joen.2020.11.021. Epub 2020 Nov 30. PMID 33271179
- [Result] Yaylali IE, Teke A, Tunca YM. The Effect of Foraminal Enlargement of Necrotic Teeth with a Continuous Rotary System on Postoperative Pain: A Randomized Controlled Trial. J Endod. 2017 Mar;43(3):359-363. doi: 10.1016/j.joen.2016.11.009. PMID 28231975
- [Result] Fazlyab M, Esmaeili Shahmirzadi S, Esnaashari E, Azizi A, Moshari AA. Effect of low-level laser therapy on postoperative pain after single-visit root canal retreatment of mandibular molars: A randomized controlled clinical trial. Int Endod J. 2021 Nov;54(11):2006-2015. doi: 10.1111/iej.13608. Epub 2021 Aug 29. PMID 34383325
- [Result] Nagendrababu V, Duncan HF, Bjorndal L, Kvist T, Priya E, Jayaraman J, Pulikkotil SJ, Pigg M, Rechenberg DK, Vaeth M, Dummer PMH. PRIRATE 2020 guidelines for reporting randomized trials in Endodontics: a consensus-based development. Int Endod J. 2020 Jun;53(6):764-773. doi: 10.1111/iej.13294. Epub 2020 Apr 23. PMID 32196696
- [Result] Nagendrababu V, Duncan HF, Bjorndal L, Kvist T, Priya E, Jayaraman J, Pulikkotil SJ, Dummer PMH. PRIRATE 2020 guidelines for reporting randomized trials in Endodontics: explanation and elaboration. Int Endod J. 2020 Jun;53(6):774-803. doi: 10.1111/iej.13304. Epub 2020 May 9. PMID 32266988
- [Result] Desai S, Chandler N. Calcium hydroxide-based root canal sealers: a review. J Endod. 2009 Apr;35(4):475-80. doi: 10.1016/j.joen.2008.11.026. Epub 2009 Feb 26. PMID 19345790
- [Result] Ruparel NB, Ruparel SB, Chen PB, Ishikawa B, Diogenes A. Direct effect of endodontic sealers on trigeminal neuronal activity. J Endod. 2014 May;40(5):683-7. doi: 10.1016/j.joen.2014.01.030. Epub 2014 Mar 20. PMID 24767564
- [Result] Zhang W, Peng B. Tissue reactions after subcutaneous and intraosseous implantation of iRoot SP, MTA and AH Plus. Dent Mater J. 2015;34(6):774-80. doi: 10.4012/dmj.2014-271. PMID 26632225
- [Result] Yoldas O, Topuz A, Isci AS, Oztunc H. Postoperative pain after endodontic retreatment: single- versus two-visit treatment. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 2004 Oct;98(4):483-7. doi: 10.1016/j.tripleo.2004.03.009. PMID 15472665
- [Result] Arslan H, Doganay E, Karatas E, Unlu MA, Ahmed HMA. Effect of Low-level Laser Therapy on Postoperative Pain after Root Canal Retreatment: A Preliminary Placebo-controlled, Triple-blind, Randomized Clinical Trial. J Endod. 2017 Nov;43(11):1765-1769. doi: 10.1016/j.joen.2017.06.028. Epub 2017 Sep 28. PMID 28967495
- [Result] Silva EJ, Menaged K, Ajuz N, Monteiro MR, Coutinho-Filho Tde S. Postoperative pain after foraminal enlargement in anterior teeth with necrosis and apical periodontitis: a prospective and randomized clinical trial. J Endod. 2013 Feb;39(2):173-6. doi: 10.1016/j.joen.2012.11.013. Epub 2012 Dec 23. PMID 23321226
- [Result] 1. Silva EJNL, Menaged K, Ajuz N, Monteiro MRFP, de Souza Coutinho-Filho T. Postoperative pain after foraminal enlargement in anterior teeth with necrosis and apical periodontitis: a prospective and randomized clinical trial. Journal of endodontics 2013;39(2):173-176. 2. Arslan H, Doğanay E, Karataş E, Ünlü MA, Ahmed HMA. Effect of low-level laser therapy on postoperative pain after root canal retreatment: a preliminary placebo-controlled, triple-blind, randomized clinical trial. Journal of endodontics 2017;43(11):1765-1769. 3. Yoldas O, Topuz A, Isçi AS, Oztunc H. Postoperative pain after endodontic retreatment: single-versus two-visit treatment. Oral Surgery, Oral Medicine, Oral Pathology, Oral Radiology, and Endodontology 2004;98(4):483-487. 4. Zhang W, Peng B. Tissue reactions after subcutaneous and intraosseous implantation of iRoot SP, MTA and AH Plus. Dental materials journal 2015;34(6):774-780. 5. Ruparel NB, Ruparel SB, Chen PB, Ishikawa B, Diogenes A. Direct effect of endodontic sealers on trigeminal neuronal activity. Journal of endodontics 2014;40(5):683-687. 6. Desai S, Chandler N. Calcium hydroxide-based root canal sealers: a review. Journal of endodontics 2009;35(4):475-480. 7. Lee B-N, Hong J-U, Kim S-M, Jang J-H, Chang H-S, Hwang Y-C, et al. Anti-inflammatory and osteogenic effects of calcium silicate-based root canal sealers. Journal of endodontics 2019;45(1):73-78. 8. Schäfer E, Bering N, Bürklein S. Selected physicochemical properties of AH Plus, EndoREZ and RealSeal SE root canal sealers. Odontology 2015;103:61-65. 9. Nagendrababu V, Duncan H, Bjørndal L, Kvist T, Priya E, Jayaraman J, et al. PRIRATE 2020 guidelines for reporting randomized trials in Endodontics: a consensus-based development. International Endodontic Journal 2020;53(6):764-773. 10. Nagendrababu V, Duncan H, Bjørndal L, Kvist T, Priya E, Jayaraman J, et al. PRIRATE 2020 guidelines for reporting randomized trials in Endodontics: explanation and elaboration. International endodontic journal 2020;53(6):774-803. 11. Fazlyab M, Esmaeili Shahmirzadi S, Esnaashari E, Azizi A, Moshari AA. Effect of low-level laser therapy on postoperative pain after single-visit root canal retreatment of mandibular molars: A randomized controlled clinical trial. International Endodontic Journal 2021;54(11):2006-2015. 12. Yaylali IE, Teke A, Tunca YM. The effect of foraminal enlargement of necrotic teeth with a continuous rotary system on postoperative pain: a randomized controlled trial. Journal of endodontics 2017;43(3):359-363. 13. Nosrat A, Dianat O, Verma P, Nixdorf DR, Law AS. Postoperative pain: an analysis on evolution of research in half-century. Journal of Endodontics 2021;47(3):358-365. 14. Gomes-Filho JE, Watanabe S, Cintra LTA, Nery MJ, Dezan-Junior E, Queiroz IOA, et al. Effect of MTA-based sealer on the healing of periapical lesions. Journal of applied oral science 2013;21(3):235-242.
- [Derived] Duzgun S, Albayrak H, Topcuoglu HS. Evaluation of the effects of calcium hydroxide-based, calcium silicate-based, and epoxy resin-based sealers on postoperative pain after a single session non-surgical endodontic retreatment: a randomized clinical trial. BMC Oral Health. 2025 Oct 9;25(1):1583. doi: 10.1186/s12903-025-06961-9. PMID 41068727